CLINICAL TRIAL: NCT05053360
Title: Effects of Healing Touch on Pain and Anxiety in Women After Cesarean
Brief Title: Healing Touch After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U20-11-4312
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative; Anxiety; Postpartum Complication
Keywords: Healing Touch
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healing Touch (Experimental): Subjects in this arm get a HT session post cesarean
  Interventions: Behavioral: Healing Touch
- Control (Active Comparator): Subjects in this arm get a control activity of equal duration
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Healing Touch — Healing Touch (HT), with a foundation in holistic nursing, is a gentle therapy that uses touch to promote health and well-being by balancing the human energy system. Healing Touch (HT) is a biofield therapy in which practitioners use their hands in a heart-centered and intentional way to provide energetic balance to support physical, emotional, mental and spiritual health. It is safe for all ages and works in harmony with, is complementary to, and may be integrated with standard medical care. Healing Touch is a collection of standardized, noninvasive techniques that clear, energize, and balance the human and
  environmental energy fields.
  Arms: Healing Touch
Other: Control — Quiet Time (QT) session is when a subject is provided with quiet for 15 minutes
  Other Names: Quiet Time
  Arms: Control

SUMMARY:
Pain and anxiety are the most common complications after cesarean birth, and impair the mother's ability to optimally care for herself and her newborn. It is important for health care providers to evaluate options post-operatively to maximize symptom management and quality of care for these patients, including the option of complementary therapies such as Healing Touch (HT). This study examines the effects of HT after cesarean delivers , including the differences between pain (Numeric Rating Scale) and anxiety (Numeric Rating scale) through a Randomized Control Trial study design. The total sample size for the proposed study will include 160 participants. The study will include patients' age ≥18 years. Based on their randomization, the study coordinator at each site will schedule either 1) a Healing Touch (HT) practitioner for the intervention group OR 2) a non-HT practitioner who will collect data for the control group. HT practitioner will verify consent, then ask the woman to complete baseline measurements of pain and anxiety. Levels of pain and anxiety will be reassessed post-intervention.

DETAILED DESCRIPTION:
Rationale: Pain and anxiety are the most common complications after cesarean birth. Pain and anxiety can impair the mother's ability to optimally care for herself and her newborn. It is important for health care providers to evaluate options post-operatively to maximize symptom management and quality of care for these patients, including the option of complementary therapies such as Healing Touch (HT).

Objectives: Primary outcomes will include the differences between the intervention and control groups' pre-/post-intervention levels of pain (Numeric Rating Scale) and anxiety (Numeric Rating scale). Secondary outcomes include the relationship between HT and demographic information of the subjects. As well, the feasibility of introducing HT as a therapy for postpartum women will be assessed.

Study Type: Randomized Control Trial

Study Design: The total sample size for the proposed study will include 160 participants. The study will include patients' age ≥18 years having a scheduled cesarean delivery at Inova Loudoun Hospital (ILH), Inova Fair Oaks Hospital (IFOH), Inova Alexandria Hospital (IAH), and Inova Fairfax Medical Campus (IFMC) who will be enrolled prior to their scheduled cesarean delivery. Inclusion criteria for the HT group are (1) the ability to ensure informed consent and completion of study assessments; (2) the ability to speak, read, and understand English; (3) scheduled cesarean delivery; (4) ≥18 years of age. Exclusion criteria for the HT group are (1) Non-English speaking due to the fidelity and variability of the research (2) Prisoners, (3) Isolation precautions, (4) active psychosis and impaired cognition, and (5) cesarean delivery who delivers prior to scheduled cesarean date. The study is expected to last about one year from study initiation through analysis.

Study Methodology: One to two weeks prior to a scheduled cesarean delivery, a member of the research team will call and screen women for eligibility on the study. If the woman electronically completes the consent form, they will be enrolled in the study and randomized into either the intervention or control group. Based on their randomization, the study coordinator at each site will schedule either 1) a Healing Touch (HT) practitioner for the intervention group OR 2) a non-HT practitioner who will collect data for the control group, and complete demographic information from the participant's medical chart. For the intervention group, the HT practitioner will verify consent, then ask the woman to complete baseline measurements of pain and anxiety. The practitioner will administer the HT intervention. Levels of pain and anxiety will be reassessed post-intervention. For the control group: a member of the research team, will ask the woman to complete baseline measurements of pain and anxiety. The subject will then be encouraged to have 15 minutes of quiet time, with the lights dimmed. After the 15 minutes of quite time, the team member will again measure the subject's levels of pain and anxiety.

Statistical Methodology: Descriptive and inferential statistical techniques will be used to determine differences between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. the ability to ensure informed consent and completion of study assessments
2. the ability to speak, read, and understand English
3. scheduled cesarean delivery
4. ≥18 years of age

Exclusion Criteria:

1. Non-English speaking due to the fidelity and variability of the research
2. Prisoners
3. Isolation precautions
4. active psychosis and impaired cognition
5. cesarean delivery who delivers prior to scheduled cesarean date -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Robinson, MSN, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Health System, Leesburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healing Touch: Subjects in this arm get a HT session post cesarean
  Healing Touch: Healing Touch (HT), with a foundation in holistic nursing, is a gentle therapy that uses touch to promote health and well-being by balancing the human energy system. Healing Touch (HT) is a biofield therapy in which practitioners use their hands in a heart-centered and intentional way to provide energetic balance to support physical, emotional, mental and spiritual health. It is safe for all ages and works in harmony with, is complementary to, and may be integrated with standard medical care. Healing Touch is a collection of standardized, noninvasive techniques that clear, energize, and balance the human and
  environmental energy fields.
Period: Overall Study
Arm/Group | Healing Touch | Control
Started | 105 | 105
Completed | 74 | 55
Not Completed | 31 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healing Touch | Control | Total
Number analyzed (Participants) | 74 | 55 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 55 | 129
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 35 [25 to 45] | 35 [25 to 45] | 35 [25 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 55 | 129
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 7 | 6 | 13
  White | 46 | 30 | 76
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants] — All participants were from the MidAtlantic region of the United States
  participants
    United States | 74 | 55 | 129

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who Reported HIGH PAIN After the Intervention
Description: Participant were asked to quantify pain using a numeric pain rating scale that range from 1 (no pain) to 10 (worst pain imaginable)
  Visual Analog Scale: Measures pain intensity. Higher scores indicate higher levels of pain 0-10 High pain = pain between 6-10 on the Visual Analog Scale
Time Frame: Immediately following intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Healing Touch | Control
Number analyzed (Participants) | 74 | 55
Participants | 2 | 7
Statistical Analysis 1: Comparison: Healing Touch vs Control; HIGH PAIN = score over 6 on a 0-10 pain scale (higher number indicating higher pain); Test type: Superiority; p = .019, Regression, Logistic; Odds Ratio (OR) = 2.87, 95% CI 2-sided [1.19 to 6.93]

2. Primary Outcome: Anxiety Measures After Intervention or Control Activity
Description: Change in anxiety before and after Healing Touch was measured using a scale with 16 questions each with a rating of 1-5, with 1=not at all and 5=extremely. The anxiety scores range from 16 to 80. Higher scores on the scale represent higher anxiety
  Hospital Anxiety Scale: Measures intensity of anxiety. Higher scores indicate higher levels of anxiety 16 Items Answer options 0-14
Time Frame: Immediately following intervention
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healing Touch | Control
Number analyzed (Participants) | 74 | 55
units on a scale | 18.8 (3.52) | 20.4 (6.4)
Statistical Analysis 1: Comparison: Healing Touch vs Control; Test type: Superiority; p = .0002, ANCOVA; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-3.47 to -1.09]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored for the duration of the study, 18 months
Arm/Group | Healing Touch | Control
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/55
Other Adverse Events (participants affected / at risk) | 0/74 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT05053360/Prot_SAP_000.pdf